CLINICAL TRIAL: NCT01536574
Title: An Open Label Extension Study With REQUIP PR for Subjects From Study ROP111528
Brief Title: Open-Label Extension Study With REQUIP PR for Subjects From Study ROP111528
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114463
Record Dates: First submitted 2012-01-19; First posted 2012-02-22 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Requip PR (Experimental): Ropinirole PR tablets of 2.0 mg, 4.0mg and 8.0 mg
  Interventions: Drug: Requip PR

INTERVENTIONS:
Drug: Requip PR — Eligible patients will be dispensed medication to uptitrate their REQUIP PR dose (2, 4, 6, 8mg respectively) during the first 4 weeks of treatment. During the 24 week treatment phase, the subjects dose will be adjusted according to the recommended schedule to achieve symptomatic control.

SUMMARY:
This open label extension study allows assessment of the long term safety profile of REQUIP PR in subjects who have completed 24 weeks of randomised treatment in study ROP111528.

Subjects must not have a break in study medication between completing the feeder study and entering extension study, treatment must be continuous.

Subjects will be dispensed down-titration medication at the study completion/early withdrawal visit and should be scheduled to return for a follow up visit 4 to 14 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have completed 24 weeks of randomised treatment in study ROP111528(and must have completed the one-week downtitration at the end of treatment/early withdrawal).
2. Subjects must not have a break in medication between completing the downtitration phase for studies ROP111528 and beginning treatment in this extension study.
3. Women of child-bearing potential must be practicing a clinically accepted method of contraception during the study and for one month following completion of the study. Acceptable contraceptive methods include oral contraception, surgical sterilization, intrauterine device (IUD), or diaphragm IN ADDITION to spermicidal foam and condom on male partner, or systemic contraception (e.g. Norplant System).
4. Provide written informed consent for this study.
5. Be willing and able to comply with study procedures.

Exclusion Criteria:

1. Patients with any ongoing clinically significant adverse events at the end of the study ROP111528.
2. Subjects with severe, clinically significant condition(s) other than Parkinson's disease which, in the opinion of the investigator, would render the subject unsuitable for the study (e.g., psychiatric, hematological, renal, hepatic, endocrinology, neurological (other than Parkinson's disease), cardiovascular, or active malignancy (other than basal cell carcinoma).
3. Subjects with clinically significant abnormalities in Laboratory or ECG tests at the end of the study ROP111528.
4. Subjects with severe dizziness or fainting due to postural hypotension on standing.
5. Withdrawal, introduction, or change in dose of hormone replacement therapy and/or any drug known to substantially inhibit CYP1A2 (e.g. ciprofloxacine, fluvoxamine, cimetidine, ethinyloestradiol) or induce CYP1A2 (e.g. tobacco, omeprazole) within 7 days prior to enrolment. Subjects already on chronic therapy with any of these agents may be enrolled but doses must have remained stable from 7 days prior to enrolment through the end of the treatment period.
6. Women who are pregnant or breast-feeding.
7. Use of an investigational drug throughout the treatment period.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2010-09-02; Primary Completion 2012-03-01 (Actual); Study Completion 2012-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- China (10):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Suzhou, Jiangsu
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Kunming, Yunnan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin

REFERENCES:
- [Derived] Zhang Z, Wang J, Zhang X, Chen S, Wang Z, Zhang B, Liu C, Qu Q, Cheng Y, Zhu R, Li J, Hu J, Cai M. An open-label extension study to evaluate the safety of ropinirole prolonged release in Chinese patients with advanced Parkinson's disease. Curr Med Res Opin. 2015 Apr;31(4):723-30. doi: 10.1185/03007995.2015.1005835. Epub 2015 Mar 12. PMID 25586298

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed 24 weeks of randomized treatment in parent Study ROP111528 (NCT01154166) and 1 week of down titration at the end of treatment or at early withdraw were allowed to enter this extension study provided they had continued on study drug without a break.
Groups:
- Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study: Participants who had received ropinirole PR in the parent double-blind (DB) study received ropinirole PR in this open-label (OL) extension study. Participants started on ropinirole PR 2 milligrams (mg) for 1 week. The dose was uptitrated weekly by 2 mg for the first 3 weeks. Later, the investigators could use their clinical judgment to increase the dose level above 8 mg once daily, in 4 mg increments, up to 24 mg once daily. Participants could remain on the same dose level if tolerability issues occurred during escalation or could reduce their dose by one dose level. After the 24-week treatment phase, all participants were down-titrated over the course of 1 week, or had an early withdraw visit if they did not complete the study for any reason. Participants returned for a follow-up visit 4-14 days after the last dose of ropinirole PR.
- Placebo in Parent DB Study, Ropinirole PR in OL Study: Participants who had received placebo in the parent DB study received ropinirole PR in this OL extension study. Participants started on ropinirole PR 2 mg for 1 week. The dose was uptitrated weekly by 2 mg for the first 3 weeks. Later, the investigators could use their clinical judgment to increase the dose level above 8 mg once daily, in 4 mg increments, up to 24 mg once daily. Participants could remain on the same dose level if tolerability issues occurred during escalation, or could reduce their dose by one dose level. After the 24-week treatment phase, all participants were down-titrated over the course of 1 week, or had an early withdraw visit if they did not complete the study for any reason. Participants returned for a follow-up visit 4-14 days after the last dose of ropinirole PR.
Period: Overall Study
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study
Started | 162 | 133
Completed | 156 | 126
Not Completed | 6 | 7
Not completed — Adverse Event | 4 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study | Total
Number analyzed (Participants) | 162 | 133 | 295
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (9.10) | 63.9 (9.87) | 64.2 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 104
  Male | 111 | 80 | 191
Race/Ethnicity, Customized [Number; unit: participants]
  Oriental | 162 | 133 | 295
Duration of Parkinson's Disease [Mean (Standard Deviation); unit: months] | 96.8 (59.68) | 105.3 (49.61) | 100.7 (55.44)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Types of Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-Treatment Phase (Comprised of the Open-label Treatment Phase and the Down-titration Phase)
Description: AE=any untoward medical occurrence (UMO), temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP. SAE=any UMO that, at any dose, results in death, is life threatening, requires hospitalization/prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomoly/birth defect. The Investigator determined if an AE/SAE was related to investigational product. Medical/scientific judgment was used to determine whether SAE reporting was appropriate in situations in which an event may not have met the SAE definition.
Time Frame: From the start of treatment (Baseline) up to Week 25
Population: Safety Population: all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study
Number analyzed (Participants) | 162 | 133
Participants
  Any AE | 58 | 56
  AE Related to Investigational Product (IP) | 33 | 35
  Any SAE | 2 | 4
  SAE Related to Investigational Product (IP) | 0 | 1
  AE Leading to Death | 0 | 0
  AE Leading to Withdrawal | 4 | 4

2. Primary Outcome: Number of Participants With the Indicated Adverse Events Related to Investigational Product During the On-treatment Phase
Description: An adverse event is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The Investigator determined if an AE/SAE was related to investigational product. The On-Treatment Phase is comprised of the Open-label Treatment Phase and the Down-titration Phase.
Time Frame: From the start of treatment (Baseline) up to Week 25
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study
Number analyzed (Participants) | 162 | 133
Participants
  Dyskinesia | 6 | 10
  Dizziness | 5 | 3
  Somnolence | 0 | 6
  Akathisia | 0 | 1
  Akinesia | 1 | 0
  Cerebral infarction | 1 | 0
  Headache | 0 | 1
  Lethargy | 0 | 1
  Syncope | 0 | 1
  Nausea | 4 | 6
  Constipation | 1 | 1
  Abdominal distension | 0 | 1
  Abdominal pain upper | 0 | 1
  Epigastric discomfort | 1 | 0
  Flatulence | 0 | 1
  Vomiting | 0 | 1
  Hallucination | 5 | 5
  Insomnia | 1 | 1
  Hallucination, auditory | 1 | 0
  Impulse-control disorder | 1 | 0
  Oedema peripheral | 1 | 1
  Gait disturbance | 1 | 0
  Medication residue | 1 | 0
  Orthostatic hypotension | 2 | 1
  Hypotension | 1 | 0
  Lymphopenia | 0 | 2
  Arrhythmia | 1 | 1
  Blood uric acid increased | 1 | 0
  Weight decreased | 1 | 0
  Muscle spasms | 1 | 0
  Musculoskeletal stiffness | 1 | 0
  Vertigo | 1 | 0
  Decreased appetite | 0 | 1
  Asphyxia | 1 | 0
  Pruritus | 0 | 1

3. Primary Outcome: Number of Participants With an Adverse Event During the Follow-up Phase
Description: as for outcome 1
Time Frame: 4- to 14-day Follow-up Phase, beginning after the date of the last dose of down-titration medication (up to and during Study Weeks 26 and 27)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study
Number analyzed (Participants) | 162 | 133
Participants
  Any AE | 2 | 3
  AE related to IP | 1 | 2
  Any SAE | 0 | 0

4. Primary Outcome: Number of Participants With the Indicated Adverse Events During the Follow-up Phase
Description: An adverse event is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. In addition to the data recorded at the follow-up visit, SAEs occurring up to and including 2 days after the last dose of down-titration medication are included in the Follow-up Phase.
Time Frame: as for outcome 3
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study
Number analyzed (Participants) | 162 | 133
Participants
  Facial palsy | 0 | 1
  Parkinsonian rest tremor | 0 | 1
  Lymphopenia | 1 | 0
  Hallucination | 0 | 1
  Choking sensation | 1 | 0

5. Primary Outcome: Number of Participants With the Indicated Adverse Events Related to Investigational Product During the Follow-up Phase
Description: An adverse event is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The Investigator determined if an AE/SAE was related to investigational product. In addition to the data recorded at the follow-up visit, SAEs occurring up to and including 2 days after the last dose of down-titration medication are included in the Follow-up Phase.
Time Frame: as for outcome 3
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study
Number analyzed (Participants) | 162 | 133
Participants
  Lymphopenia | 1 | 0
  Parkinsonian rest tremor | 0 | 1
  Hallucination | 0 | 1

6. Secondary Outcome: Mean Gambling Symptom Assessment Scale (G-SAS) Score at Week 24
Description: The G-SAS is a reliable and valid self-reported measure of gambling symptoms. It is comprised of twelve questions aimed at evaluating gambling symptoms; each item is scored on a 5-point scale from 0 (no symptoms) to 4 (extreme symptoms). The total score ranges from 0 to 48, where 0=least severe and 48=most severe.
Time Frame: Week 24
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed. Data were collected using the last observation carried forward (LOCF) method: the last available on-therapy observation for a participant was used to estimate missing data points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study
Number analyzed (Participants) | 158 | 129
Scores on a scale | 0.9 (4.03) | 1.3 (4.32)

7. Secondary Outcome: Mean Change From Baseline in the Gambling Symptom Assessment Scale (G-SAS) Score at Week 24
Description: The G-SAS is a reliable and valid self-reported measure of gambling symptoms. It is comprised of twelve questions aimed at evaluating gambling symptoms; each item is scored on a 5-point scale from 0 (no symptoms) to 4 (extreme symptoms). The total score ranges from 0 to 48, where 0=least severe and 48=most severe. Change from Baseline is calculated as the value at Week 24 minus the Baseline value.
Time Frame: Baseline and Week 24
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed. Data were collected using the LOCF method.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study
Number analyzed (Participants) | 158 | 129
Scores on a scale | -0.1 (2.87) | -0.3 (4.64)

ADVERSE EVENTS:
Time Frame: AEs and SAEs are presented for the On-treatment Phase, including the Open-label Treatment Phase (24 weeks) and the Down-titration Phase (1 week) (up to Study Week 25).
Arm/Group | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study | Placebo in Parent DB Study, Ropinirole PR in OL Study
Serious Adverse Events (participants affected / at risk) | 2/162 | 4/133
Other Adverse Events (participants affected / at risk) | 58/162 | 56/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study (N=162) | Placebo in Parent DB Study, Ropinirole PR in OL Study (N=133)
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Retinal hemorrhage (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole PR in Parent DB Study, Ropinirole PR in OL Study (N=162) | Placebo in Parent DB Study, Ropinirole PR in OL Study (N=133)
Dyskinesia (Nervous system disorders) | 7 | 11
Dizziness (Nervous system disorders) | 7 | 5
Somnolence (Nervous system disorders) | 2 | 6
Headache (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 2
Akathisia (Nervous system disorders) | 0 | 1
Akinesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Cerebral disorder (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischemia (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Meralgia paraesthetica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 5 | 5
Sleep disorder (Psychiatric disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 2 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0
Impulse-control disorder (Psychiatric disorders) | 1 | 0
Weight decreased (Investigations) | 3 | 4
Weight increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 2 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Edema peripheral (General disorders) | 1 | 2
Chest discomfort (General disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Medication residue (General disorders) | 1 | 0
Edema (General disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Retinal hemorrhage (Eye disorders) | 1 | 0
Hypersensitvity (Immune system disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.